CLINICAL TRIAL: NCT03949075
Title: Impact of Angiotensin Converting Enzyme Activity on Exercise Training Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18016341
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Exercise; Angiotensin-Converting Enzyme Inhibitors
Keywords: Adaptation, Physiological; Genotype; Polymorphism, Genetic; Enalapril; Physiological Effects of Drugs
MeSH Terms: conditions — Motor Activity | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The present study is double-blinded with regard to ACE genotype and study medication and the blinding is kept until completion of the trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enalapril treatment (Experimental)
  Interventions: Drug: Enalapril
- Placebo treatment (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enalapril — Participants will be assigned to daily administration of ACE inhibitors (Initially 5 mg Corodil® 'Enalapril' daily followed by up to 20 mg daily dependent on the blood pressure response) combined with an 8-week training period.
  Arms: Enalapril treatment
Drug: Placebo — Participants will be assigned to daily administration of placebo (5-20 mg CaCO3) combined with an 8-week training period.
  Arms: Placebo treatment

SUMMARY:
The phenotype based on the insertion/deletion (I/D) polymorphism of the human angiotensin converting enzyme (ACE) gene has been associated with individual training response. Briefly, intervention studies have demonstrated an 11-fold greater training-induced improvement in muscular endurance for ACE I/I homozygotes compared to ACE D/D homozygotes.

Importantly, the ACE I/D polymorphism causes large inter-individual differences in serum ACE activity. Because the ACE D/D genotype is characterized by high plasma ACE activity and potentially blunted endurance exercise training response, it appears likely that ACE inhibitors (ACEi) have the potential to improve the outcome of exercise training for ACE D/D homozygotes.

Thus, in the present study the investigators apply a randomized double-blind placebo-controlled longitudinal design to investigate whether pharmacological inhibition of ACE activity can amplify the exercise training response in healthy humans carrying either the ACE D/D or ACE I/I genotype.

The study hypothesis is that inhibition of ACE activity in healthy humans with the ACE D/D genotype will amplify the health beneficial effects of exercise training while this is not the case in ACE I/I homozygotes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-50 years
* Healthy

Exclusion Criteria:

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Maximal systemic oxygen uptake | 20 minutes
  Training-induced changes in maximal systemic oxygen uptake (L/min) is evaluated with an incremental maximal cycle protocol on a cycle ergometer
Skeletal muscle endurance | 5 minutes
  Training-induced changes in muscle endurance evaluated as changes in duration (sec) of a repetitive elbow-flexion exercise

SECONDARY OUTCOMES:
Blood volume | 20 minutes
  Training-induced changes in total blood volume (mL) is measured using the Carbon-monoxide rebreathing method.
Endurance performance | 15 minutes
  Training-induced changes in endurance performance is determined by a 2000 meter time trial on an indoor rowing ergometer
Skeletal muscle oxidative capacity | 60 minutes
  Training-induced changes in muscle oxidative capacity is evaluated as maximal citrate synthase and 3- hydroxy-acetylCoa-dehydrogenase activity (µmol/g/min)
Mitochondrial biogenesis | 60 minutes
  Expression of complex I-V will be analyzed in order to evaluate if the applied training induced mitochondrial biogenesis.
Mean arterial pressure (MAP) | 10 minutes
  Training-induced changes in resting MAP (mmHg) will be estimated using this formula: MAP = diastolic pressure + 1/3 (systolic pressure - diastolic pressure)
Steady-state systemic oxygen uptake | 10 minutes
  Training-induced changes in steady-state systemic oxygen uptake (mL/min) is determined by indirect calorimetry during a submaximal cycle protocol on a cycle ergometer
Muscle strength | 1 minute
  Training-induced changes in muscle strength (kg) is measured using a handgrip dynamometer
Fat mass | 20 minutes
  Training-induced changes in fat mass (kg) is determined by dual-energy x-ray absorptiometry (DXA)-scan
Fat free mass | 20 minutes
  Training-induced changes in fat free mass (kg) is determined by DXA-scan
Body fat percentage | 20 minutes
  Training-induced changes in body fat percentage (%) is determined by DXA-scan
Left ventricular (LV) mass | 45 minutes
  Training-induced changes in LV mass (g) is determined by cardiac magnetic resonance imaging (cMRI)
LV end-diastolic volume | 45 minutes
  Training-induced changes in LV end-diastolic volume (mL) is determined by cMRI
LV mean wall thickness | 45 minutes
  Training-induced changes in LV mean wall thickness (cm) is determined by cMRI
LV stroke volume | 45 minutes
  Training-induced changes in LV stroke volume (mL) is determined by cMRI
LV ejection fraction | 45 minutes
  LV stroke volume (mL) and LV end-diastolic volume (mL) will be used to measure training-induced changes in LV ejection fraction (%)

OTHER OUTCOMES:
ACE activity | 10 minutes
  Obtained blood samples will be analyzed for ACE activity

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai B Nordsborg, phD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymous data will be shared with other researchers.

REFERENCES:
- [Background] Rigat B, Hubert C, Alhenc-Gelas F, Cambien F, Corvol P, Soubrier F. An insertion/deletion polymorphism in the angiotensin I-converting enzyme gene accounting for half the variance of serum enzyme levels. J Clin Invest. 1990 Oct;86(4):1343-6. doi: 10.1172/JCI114844. PMID 1976655
- [Background] Montgomery HE, Marshall R, Hemingway H, Myerson S, Clarkson P, Dollery C, Hayward M, Holliman DE, Jubb M, World M, Thomas EL, Brynes AE, Saeed N, Barnard M, Bell JD, Prasad K, Rayson M, Talmud PJ, Humphries SE. Human gene for physical performance. Nature. 1998 May 21;393(6682):221-2. doi: 10.1038/30374. No abstract available. PMID 9607758
- [Derived] Sjuretharson T, Bejder J, Breenfeldt Andersen A, Bonne TC, Kyhl K, Thomassen M, Prats J, Oddmarsdottir Gregersen N, Skoradal MB, Weihe P, Nordsborg NB, Mohr M. Robust arm and leg muscle adaptation to training despite ACE inhibition: a randomized placebo-controlled trial. Eur J Appl Physiol. 2023 Feb;123(2):325-337. doi: 10.1007/s00421-022-05072-5. Epub 2022 Oct 22. PMID 36271942